CLINICAL TRIAL: NCT05403892
Title: Inter and Intra-observer Reliability and Validity of the Ankle Dorsiflexion Lunge Test With a Level Laser in Healthy Teenage Athletes: a Novel Way of Measuring.
Brief Title: Reliability and Validity of a New Ankle Dorsiflexion Lunge Test Using a Level Laser.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Ballardin Francesco, Clinical Professor, University of Bologna
Other Study IDs: TMUNIBO2022TT
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Ankle Joint; Range of Motion, Articular; Reliability and Validity
Keywords: level laser; dorsiflexion lunge test; ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant: The participants must be teenage basketball players (12-17 years old).
  The exclusion criteria are:
  * have suffered in the last 3 months of lower limb musculoskeletal disorders such as pain for more than 7 days (ankle distortion outcomes, leg/foot fractures, plantar heel pain, metatarsalgias, etc);
  * athletes who have undergone surgery on their lower limb.
  Interventions: Diagnostic Test: level laser lunge test; Diagnostic Test: dorsiflexion Lunge test

INTERVENTIONS:
Diagnostic Test: level laser lunge test — In order to perform the Level Laser Test, the operator 1 places a laser lever on the ground one metre aside and 50 cm forward the ankle to be examined. This laser (a 2-class laser not harmful to the eyes) maintains a linear laser light beam perpendicular to the floor. The examined leg is placed further forward to the other one, as it happens in the DLT. The teenage performs a forward lunge perpendicularly to the laser line, the heel positioning 50 cm from the laser line. Operator 1 has the subject perform a lunge while operator 2 measures the distance from the kneecap to the laser line. The measurement, deducted by 50 cm, leads to the heel-to-wall distance (value used to DLT).
Diagnostic Test: dorsiflexion Lunge test — The dorsiflexion lunge test (DLT) will be used to measure ankle dorsiflexion. To perform this test, the teenage stands in front of a wall holding the foot of their limb to be measured perpendicularly to it. The other foot is to be kept behind it. The teenage is asked to perform a lunge (to dorsiflex the ankle and bring the knee into flexion) until the front knee touches the wall without the heel lifting off the ground. The teenage steps away from the wall as much as possible as long as the knee keeps touching the wall. Measurement in centimeters is taken from the heel of the examined leg to the wall.
  Other Names: weight bearing lunge test

SUMMARY:
The study aims to find validity and intra-inter examiner reliability of the Lever Laser Lunge Test (LLLT). This is a new way to measure ankle range of motion during weight bearing, instead of classical dorsiflexion lunge test The study wants to assume that LLLT is comparable to the traditional test but more efficient because it could be used in different settings.

To reach this goal, these two non-invasive tests will be performed to measure the amount of movement of the ankle joint in healthy teenage basketball players.

Data will be statistically compared and studied.

DETAILED DESCRIPTION:
The dorsiflexion lunge test or knee-to-wall test (DLT) measure the range of movement of weight bearing ankle dorsiflexion. This test is frequently used in sport setting, in order to identify ankle limitations which could lead to possible injuries or joint overloads.

DLT is a cheap and simple measurement method to assess the ankle dorsiflexion, however clinicians find possible bias that reduce the usability of this test.

In order to remove this bias, this study suggests a new measurement method carried out by a level laser to create a virtual wall (the vertical red line produced by the laser).

The study aims therefore to estimate the validity and intra-inter examiner reliability of this method, in comparison to the DLT.

The instruments used are a professional level laser and a rigid ruler. A group of male teenager basketball players from Bologna competitive sports clubs will be recruited.

In order to assess the validity of this new test the clinicians will compare statistically the outcome of both test In order to assess the intra and inter examiner reliability the clinicians will compare repeated measurements of the LLLT.

It is assumed that both measurement methods (traditional and laser method) have comparable validity but LLLT reliability intra and inter examiner should be higher than the DLT one.

ELIGIBILITY:
Inclusion Criteria:

* male teenagers basketball players enrolled in a competitive sports club;
* teenagers whose parents have signed the privacy and consent forms.

Exclusion Criteria:

* athletes who have suffered in the last 3 months of lower limb musculoskeletal disorders such as pain for more than 7 days (ankle distortion outcomes, leg/foot fractures, plantar heel pain, metatarsalgias, etc);
* athletes who have undergone surgery on their lower limb.

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Male teenagers basketball players from Bologna competitive sports clubs.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-28 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
validity of lever laser lunge test | 1 day
  the collected values will be statistically processed to identify a significant validity of the LLLT comparing to the DLT
intra-examiner reliability of lever laser lunge test | 2 days
  the collected values will be statistically processed to identify a significant intra-examiner reliability of the LLLT compared to the DLT values found in the bibliography
inter-examiner reliability of lever laser lunge test | 2 days
  the collected values will be statistically processed to identify a significant inter-examiner reliability of the LLLT compared to the DLT values found in the bibliography

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Torriglia, Principal Investigator — Università degli studi di Bologna; Pillastrini Paolo, Study Director — Università degli studi di Bologna; Silvia Pozzan, Study Chair — Università degli studi di Bologna
Locations (1):
- Dipartimento di Scienze Biomediche e Neuromotorie (DIBINEM), Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be sharing by a publication and will be stored and shared with those who request it while maintaining the anonymity of participants.

REFERENCES:
- [Background] Hall EA, Docherty CL. Validity of clinical outcome measures to evaluate ankle range of motion during the weight-bearing lunge test. J Sci Med Sport. 2017 Jul;20(7):618-621. doi: 10.1016/j.jsams.2016.11.001. Epub 2016 Nov 23. PMID 28108266
- [Background] Kang MH, Oh JS. Relationship Between Weightbearing Ankle Dorsiflexion Passive Range of Motion and Ankle Kinematics During Gait. J Am Podiatr Med Assoc. 2017 Jan;107(1):39-45. doi: 10.7547/14-112. PMID 28271931
- [Background] Konor MM, Morton S, Eckerson JM, Grindstaff TL. Reliability of three measures of ankle dorsiflexion range of motion. Int J Sports Phys Ther. 2012 Jun;7(3):279-87. PMID 22666642
- [Background] Munteanu SE, Strawhorn AB, Landorf KB, Bird AR, Murley GS. A weightbearing technique for the measurement of ankle joint dorsiflexion with the knee extended is reliable. J Sci Med Sport. 2009 Jan;12(1):54-9. doi: 10.1016/j.jsams.2007.06.009. Epub 2007 Sep 20. PMID 17888733
- [Background] Rose KJ, Burns J, North KN. Factors associated with foot and ankle strength in healthy preschool-age children and age-matched cases of Charcot-Marie-Tooth disease type 1A. J Child Neurol. 2010 Apr;25(4):463-8. doi: 10.1177/0883073809340698. Epub 2009 Aug 11. PMID 19671887
- [Result] Bennell KL, Talbot RC, Wajswelner H, Techovanich W, Kelly DH, Hall AJ. Intra-rater and inter-rater reliability of a weight-bearing lunge measure of ankle dorsiflexion. Aust J Physiother. 1998;44(3):175-180. doi: 10.1016/s0004-9514(14)60377-9. PMID 11676731
- [Result] Cejudo A, Sainz de Baranda P, Ayala F, Santonja F. A simplified version of the weight-bearing ankle lunge test: description and test-retest reliability. Man Ther. 2014 Aug;19(4):355-9. doi: 10.1016/j.math.2014.03.008. Epub 2014 Apr 2. PMID 24746162
- [Result] Gatt A, Chockalingam N. Clinical assessment of ankle joint dorsiflexion: a review of measurement techniques. J Am Podiatr Med Assoc. 2011 Jan-Feb;101(1):59-69. doi: 10.7547/1010059. PMID 21242472
- [Result] Langarika-Rocafort A, Emparanza JI, Aramendi JF, Castellano J, Calleja-Gonzalez J. Intra-rater reliability and agreement of various methods of measurement to assess dorsiflexion in the Weight Bearing Dorsiflexion Lunge Test (WBLT) among female athletes. Phys Ther Sport. 2017 Jan;23:37-44. doi: 10.1016/j.ptsp.2016.06.010. Epub 2016 Jun 29. PMID 27665249
- [Result] Powden CJ, Hoch JM, Hoch MC. Reliability and minimal detectable change of the weight-bearing lunge test: A systematic review. Man Ther. 2015 Aug;20(4):524-32. doi: 10.1016/j.math.2015.01.004. Epub 2015 Jan 29. PMID 25704110
- See also: A study to determine the reliability of an ankle dorsiflexion weight-bearing device — https://doi.org/10.1016/j.physio.2005.04.005